CLINICAL TRIAL: NCT03233594
Title: PET Imaging of Chronic Pain Syndromes
Status: Active, not recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 17D.163
Record Dates: First submitted 2017-06-29; First posted 2017-07-28 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain Syndrome
Keywords: Chronic Pain Syndrome; Chronic Pain; Chiropractic; PET; MRI; Positron emission tomography; Magnetic resonance imaging; Neuro Emotive Technique (NET)
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chiropractic Group: Participants receiving a chiropractic care technique Neuro Emotive Technique (NET) will complete initial pain evaluations and questionnaires for chronic pain symptoms. After approximately 8 weeks participants will receive follow evaluation for pain. Pre and Post PET-MRI scan will be conducted to evaluate changes.
  Interventions: Other: Chiropractic Group
- Healthy Control Group: Participants will receive initial evaluations and questionnaires followed by a PET-MRI scan.
  Interventions: Other: Healthy Control Group

INTERVENTIONS:
Other: Chiropractic Group — Participants will receive approximately 8 weeks of chiropractic care.
  Groups: Chiropractic Group
Other: Healthy Control Group — Participants will not receive any interventions.
  Groups: Healthy Control Group

SUMMARY:
Central nervous system (CNS) changes associated with pain have been difficult to measure until the development of functional neuroimaging techniques such as positron emission tomography (PET). We have previously observed asymmetry in the thalamus associated with chronic pain that altered during acupuncture therapy. Imaging studies of therapeutic techniques for chronic pain in animals and humans have been quite limited. This study will be the first to utilize FDG PET-MRI imaging of both the brain and body in order to assess CNS changes and peripheral body changes related to chronic pain and its potential management.

DETAILED DESCRIPTION:
The proposed study is based on our growing understanding of chronic pain and our ability to use functional brain imaging to study in vivo neurophysiologic processes. It is important to understand the brain and body mechanisms of chronic pain in order to better determine therapeutic interventions to reduce pain. Part of the difficulty in treating chronic pain is to determine how better to diagnose what specific issues are affecting the brain and body that result in chronic pain. Participants will undergo a small battery of diagnostic tests that include magnetic resonance imaging (MRI), positron emission tomography (PET). A secondary goal of this study is to determine if undergoing chiropractic care alters body or brain physiology in patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria for Chronic Pain Patients:

* Age greater than 18 years old.
* Have chronic pain symptoms for >3 months;
* Have moderate pain (>3/10) in 2 or more areas for more than 5 out of 7 days
* Is planning on undergoing chiropractic care for the clinical management of the chronic pain.
* May be on pain medications provided that they are on a stable dose for at least 1 month
* Patients have no other pre-existing and active significant medical, neurological, or psychological disorders.
* Minor, stable health problems that should have no substantial effect on cerebral blood flow will be allowed (i.e. controlled hypertension, medication controlled diabetes).
* Patients will be allowed to be taking medications or supplements at the initial intake, but they must be on a stable dose regimen for at least 1 month.
* Able to give informed consent and willing to complete the study at Thomas Jefferson University and Marcus Institute of Integrative Health.

Inclusion Criteria for Healthy Controls:

* No significant current active medical conditions.
* Stable medical conditions as determined by the PI are allowed.
* No brain or body abnormalities that would affect the acquisition or analysis of the scan.

Exclusion Criteria for Chronic Pain Patients and Healthy Controls:

* Pregnant or breast feeding
* Enrollment in active clinical trial/ experimental therapy within the prior 30 days.
* Subject is unable or unwilling to lie still in the scanner (i.e. due to claustrophobia or weight)
* Subject has metal in their body or other reason that they cannot undergo magnetic resonance imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited only if they are already planning on receiving standard clinical chiropractic care for their pain.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Use combined PET/MRI to define pain activity pattern and inflammation. | Baseline and 8 weeks
  To use PET-MRI to define abnormal brain and body activity and evaluate changes in inflammation in painful regions in patients with chronic pain syndromes.

SECONDARY OUTCOMES:
Use combined PET/MRI to demonstrate brain and body activity in responders and non-responders. | Baseline and 8 weeks
  Patterns will be compared between those who respond and those who do not respond to chiropractic care.

OTHER OUTCOMES:
Brief Pain Inventory Questionnaire | Baseline and 8 weeks
  This validated questionnaire will be used as one of the evaluation questionnaires for the study.
Numeric Rating Scale for Pain Intensity for specific locations | Baseline and 8 weeks
  This validated questionnaire will be used as one of the evaluation questionnaires for the study.
Profile of Mood Scale | Baseline and 8 weeks
  The Profile of Mood States (POMS) is a validated questionnaire of 65 single word items that asks "How have you been feeling in the past week including today." The subjects will select their response to each word that describes a mood or feeling on a Likert scale from 1= Not at All, 2= A Little, 3=Moderately, 4=Quite a lot, to 5=Extremely. The responses are scored to generate values for Tension, Anger, Confusion, Depression and Vigor. The higher scores indicate a greater presence of that mood or state.
Patient-Reported Outcomes Measurement Information System (PROMIS) for quality of life assessment | Baseline and 8 weeks
  This validated questionnaire will be used as one of the evaluation questionnaires for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B. Newberg, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Villanova, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT03233594/ICF_005.pdf